CLINICAL TRIAL: NCT01132053
Title: Role of Inflammation in PML
Brief Title: Role of Inflammation in Progressive Multifocal Leukoencephalopathy (PML)
Status: Completed | Type: Observational
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Chen Sabrina Tan, principal investigator, Beth Israel Deaconess Medical Center
Other Study IDs: 2004P000089; NS 047029 (Other Grant/Funding Number: NIH)
Record Dates: First submitted 2010-05-26; First posted 2010-05-27 (Estimated); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Progressive Multifocal Leukoencephalopathy
Keywords: JC Virus
MeSH Terms: conditions — Leukoencephalopathy, Progressive Multifocal

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, Urine, CSF if needed for clinical management.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- PML: These are subjects who have confirmed PML.
- Control: These are subjects who do not have PML. They may be healthy or immune compromised due to Cancer, Transplant, or HIV.

SUMMARY:
This is a continuation of our previous studies on Progressive Multifocal Leukoencephalopathy (PML). We will focus on the role of inflammation in PML, and define prognostic markers of disease evolution.

DETAILED DESCRIPTION:
To determine precisely what are the host or viral factors that may predict a favorable outcome for PML patients and the role of inflammation in preventing JCV from causing brain disease. One of the goals of this study is to help establish non-invasive markers of PML evolution by studying the brain metabolism in PML lesions using Magnetic Resonance Imaging (MRI), Magnetic Spectroscopy (MRS) and other advanced imaging modalities.

ELIGIBILITY:
Inclusion Criteria:

* PML patients of 18 years of age or older will be included in this study.

Exclusion Criteria:

1. Presence of opportunistic brain lesions other than PML. ( e.g., toxoplasmosis, lymphoma)
2. Presence of confounding neurological disorder such as brain neoplasm etc.

In addition patients with a contraindication to MRI examination will be excluded from study. Contraindications to the MRI examination include:

1. Medically unstable or hematological, renal, or hepatic dysfunction.
2. Cardiac pacemaker
3. Internal clips,
4. Metal implants, or external clips with 10 mm of the head.
5. Metal in the eyes.
6. Pregnant
7. Claustrophobia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: PML patients of 18 years of age or older in the Boston area will be included in this study.
  The control groups will include HIV+ and HIV- individuals who need to have a lumbar puncture for their clinical management.
Sampling Method: Non-Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2004-06 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chen S Tan, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

REFERENCES:
- See also: Description of PML studies at BIDMC — http://bidmc.org/CentersandDepartments/Departments/Neurology/HIVNeurologyClinic/ClinicalStudies.aspx